CLINICAL TRIAL: NCT03243266
Title: DxH520 Pediatric Reference Interval Verification
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: B90590
Record Dates: First submitted 2017-07-28; First posted 2017-08-08 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- CBC/Diff Reference Interval: Hematology routine diagnostic test
  Interventions: Diagnostic Test: CBC/Diff Reference Interval

INTERVENTIONS:
Diagnostic Test: CBC/Diff Reference Interval — Results will not be used to manage patients

SUMMARY:
Results from this study will be used to verify that the published pediatric reference intervals are met on the DxH 520 Hematology Analyzer for the pediatric age ranges.

DETAILED DESCRIPTION:
Pediatric specimens from each age range will be tested from apparently healthy children. Ten male and Ten female are required for each age range. The values will be assessed against published reference ranges to verify that the values obtained fall within the expected reference interval for the age ranges listed below:

1. Neonate: 0 to 30 days
2. Infant: > 30 days to 2 years
3. Child: 3 years to 12 years
4. Adolescent: 13 years to 21 years

ELIGIBILITY:
Inclusion Criteria:

* All subject genders, race and ethnicity will be included in the study. Pediatric samples will be targeted for this study within the specified age ranges.
* Specimens should be from apparently healthy individuals.
* Samples from inpatient and ED visits maybe included if they are confirmed to be the final CBC before discharge and the patient had a non-hematological diagnosis

Exclusion Criteria:

* Samples originating from a hematology/oncology clinic (both inpatient and outpatient)
* Samples originating from a patient with a hematological disorder or diagnosis
* Samples from the Neonatal Intensive Care Unit that are not the last specimens collected prior to discharge

Ages: 1 Minute to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male, Female
Study Population: Pediatric specimens from apparently healthy children
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Pediatric Reference Interval Verification of Hematology CBC/Diff parameters | 1 day
  Verify Reference Intervals of Hematology CBC/Diff parameters in pediatric age groups. The blood cell count test parameters to be verified are:
  White Blood Cells (x10^3/µL), Red Blood Cells (x10^6/µL), Hemoglobin (g/dL), Hematocrit %, Mean Corpuscular Hemoglobin (pg), Mean Corpuscular Hemoglobin Concentration (g/dL), Mean Corpuscular Volume (fL), Red Cell Distribution Width-CV (%) Red cell Distribution Width-SD (fL), Platelets (x10^3/µL), Mean Platelet Volume (fL), Neutrophil %, Neutrophil Count (x10^3/µL), Lymphocyte %, Lymphocyte Count (x10^3/µL), Monocyte %, Monocyte Count (x10^3/µL), Eosinophil %, Eosinophil Count (x10^3/µL), Basophil %, Basophil Count (x10^3/µL). Study results will be analyzed following CLSI guideline EP28-A3c.

CONTACTS AND LOCATIONS:
Overall Officials: Khosrow Adeli, Ph.D, Principal Investigator — The Hospital for Sick Children; Meer-Taher Shabani-Rad, MD, Principal Investigator — Alberta Children's Hospital
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario